CLINICAL TRIAL: NCT02568202
Title: Bridging Hemophilia B Experiences, Results and Opportunities Into Solutions (B-HERO-S)
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: HAEM-4268; U1111-1171-8168 (Other: WHO)
Record Dates: First submitted 2015-09-18; First posted 2015-10-05 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Haemostasis; Congenital Bleeding Disorder; Haemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — This is an online web-based cross-sectional survey in which participants will complete one of two questionnaires.
  There will be no treatment.

SUMMARY:
This study is conducted in the United States of America (USA). Tha aim of this study is bridging Hemophilia B Experiences, Results and Opportunities into Solutions (B-HERO-S).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged below or equal to 18 years with hemophilia B (any severity, with or without inhibitors)
* Caregivers of children currently aged below 18 years with hemophilia B (any severity, with or without inhibitors)
* Subjects must have access to the internet, either at home or at a location convenient to them
* Provision of informed consent before the start of any survey-related activities

Exclusion Criteria:

* Inability to understand and comply with written instructions in English
* Previous completion of the B-HERO-S study with receipt of compensation
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will investigate adult patients at least 18 years of age with mild-severe hemophilia B and caregivers of children (current age below 18 years) with hemophilia B.
Sampling Method: Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
An online survey of Prevalence and characteristics of adults with hemophilia B | At day 0
An online survey of Prevalence and characteristics of children with hemophilia B (and their parents) | At day 0
An online survey of Prevalence of psychosocial and other comorbidities in patients with hemophilia B | At day 0

SECONDARY OUTCOMES:
Percentage of participants reporting difficulty with access to treatment (e.g. factor) | At day 0
An online survey of Percentage of participants reporting difficulty with access to treatment centers | At day 0
Percentage of participants reporting hemophilia interference with employment/education | At day 0
Percentage of participants reporting hemophilia interference with physical activities | At day 0
Percentage of participants reporting hemophilia interference with relationships | At day 0
Health related quality of life: EuroQol | At day 0
Health related quality of life:EQ-5D-5L | At day 0
Health related quality of life: VAS (Visual Analog Scale) | At day 0
Health related quality of life: BPI (Brief Pain Inventory) short form - Pain severity and interference | At day 0
Health related quality of life: HAL (Hemophilia Activities List) | At day 0
Health related quality of life: HemoCAB (Caregiver Hemophilia Burden Scale | At day 0
Drivers of psychosocial impact (e.g. hemophilia severity, age, weight, prior treatment history, education) | At day 0

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Plainsboro, New Jersey, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com